CLINICAL TRIAL: NCT00838708
Title: A Phase II, Randomised, Double-blind, Vehicle-controlled, Cross-over Study to Determine the Anti-pruritic Efficacy, Safety and Local Dermal Toleration of SRD174 Cream in Subjects With Atopic Dermatitis.
Brief Title: Phase IIa Safety and Efficacy Study of SRD174 Cream in Patients With AD-associated Pruritus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Serentis Ltd. (Industry)
Responsible Party: Robert Tansley, Chief Medical Officer, Serentis
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P174954201CD
Record Dates: First submitted 2009-02-05; First posted 2009-02-06 (Estimated); Last update posted 2009-10-30 (Estimated); Status verified 2009-10

CONDITIONS: Pruritus, Atopic Dermatitis
MeSH Terms: conditions — Pruritus; Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vehicle cream (Placebo Comparator)
  Interventions: Other: vehicle cream
- SRD174 Cream (Experimental)
  Interventions: Drug: SRD174 Cream

INTERVENTIONS:
Drug: SRD174 Cream — topical SRD174 Cream
  Arms: SRD174 Cream
Other: vehicle cream — topical vehicle cream
  Arms: Vehicle cream

SUMMARY:
Pruritus is an essential feature for the diagnosis of atopic dermatitis and may play an important part in disease progression. Itching has a significant impact on the quality of life of AD sufferers, in particular night-time itching leading to sleep disturbance and subsequent poor daytime performance.

The objective of this study is to determine whether SRD174 Cream is a safe and effective therapy for moderate to severe pruritus associated with atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18 years and over moderate to severe AD pruritus
* Written signed and dated informed consent
* Satisfactory medical assessment with no clinically relevant abnormalities

Exclusion Criteria:

* Subject with active and pruritic AD covering a body surface area (BSA) > 20%
* Subject with severe AD defined as an IGA score of 4
* Subject with current or recurrent skin disease (except AD) that could affect the site of application of action, absorption or disposition of the investigational product, or clinical, laboratory assessments.
* Subjects with unstable or uncontrolled medical conditions that could require intensive treatment during the course of the study.
* Subject with known or suspected intolerance or hypersensitivity to the Investigational products or any of the stated ingredients.
* Subject who has a medical or psychiatric condition or laboratory abnormality that may increase the risk associated with trial participation or investigational product administration or may interfere with interpretation of trial results and, in the judgment if the investigator, would make the subject inappropriate for entry into this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2009-01; Primary Completion 2009-07 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Measure of intensity and duration of itch episodes | Duration of episode

SECONDARY OUTCOMES:
Safety and local dermal tolerability | 4 weeks

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Birmingham, Alabama
  - Hot Springs, Arkansas
  - Oceanside, California
  - Ormond Beach, Florida
  - Detroit, Michigan
  - Grand Blanc, Michigan
  - High Point, North Carolina
  - Winston-Salem, North Carolina
  - Hazleton, Pennsylvania
  - Philadelphia, Pennsylvania
  - Dallas, Texas
  - Lynchburg, Virginia
  - Spokane, Washington